CLINICAL TRIAL: NCT05500677
Title: Comparison of the Analgesic Efficacy of Lidocaine Spray Versus Tramadol and Fentanyl for Pain Control in Rib Fractures: A Prospective, Randomized, Controlled and Open-label Study
Brief Title: Lidocaine Spray for Pain Control in Rib Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ahmet Burak Erdem, M.D., Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Record Dates: First submitted 2022-07-29; First posted 2022-08-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Rib Fractures; Analgesia
Keywords: Analgesia; Fentanyl; Lidocaine spray; Rib fracture; Tramadol
MeSH Terms: conditions — Rib Fractures; Agnosia | interventions — Lidocaine; Tramadol; Fentanyl

STUDY DESIGN:
Intervention Model Description: Pain control in rib fracture
Masking Description: open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine (Active Comparator): 10% lidocaine spray was applied on the broken rib from a distance of 10 cm, 1-2 puffs. Each puff contains 10 mg of lidocaine.
  Interventions: Drug: Lidocaine topical
- Tramadol (Active Comparator): 100 mg of tramadol hydrochloride was placed in 150 cc isotonic saline and given as a 15-minute intravenous infusion.
  Interventions: Drug: Lidocaine topical
- Fentanyl (Active Comparator): 50 mcg of fentanyl citrate was given as a 15-minute intravenous infusion in 150 cc isotonic.
  Interventions: Drug: Lidocaine topical

INTERVENTIONS:
Drug: Lidocaine topical — Lidocaine spray, which is a quick and easy-to-use topical local anesthetic, will be applied as a puff to the painful area.
  Other Names: Tramadol hydrochloride; Fentanyl citrate

SUMMARY:
In this study, we aimed to compare the analgesic efficacy of lidocaine spray with tramadol hydrochloride and fentanyl citrate in rib fractures.

DETAILED DESCRIPTION:
Patients over the age of 18 who came to our emergency department with blunt chest trauma were divided into three groups. Groups was created from patients who were given lidocaine 10% spray (local), i.v. 100 mg of tramadol and i.v. fentanyl 50 mcg. A total of 48 patients, each of whom were 16, were included in the study. Numerical rating scale (NRS) pain scores of the patients at baseline, 15th, 30th and 60th minutes were compared. These scores and the amount of falls at follow-up were analyzed comparatively between the 3 groups.

ELIGIBILITY:
Inclusion Criteria:

* Open conscious
* Oriented and cooperative
* Blunt thoracic trauma and rib fracture
* Numerical rating scale (NRS) was 5 or higher

Exclusion Criteria:

* Patients who refused to participate in the study
* Detected or suspected pregnancy
* Known history of allergy or other adverse reaction to the drugs used in the study
* History of sedative drug use or drug addiction
* Analgesic use within 6 hours of admission to the emergency department
* Needed emergency tube thoracostomy or surgical intervention
* Hemodynamically unstable
* Open and/or infected wounds in the fracture area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Pain control | 60th minutes.
  We use Numeric rating scala.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Burak Erdem, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No